CLINICAL TRIAL: NCT07020455
Title: Is The Combine Prolotherapy More Effective Than The Traditional Prolotherapy In Patients With Temporomandibular Joint Hypermobility?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Halenur Ateş, DDS, Karadeniz Technical University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025/6
Record Dates: First submitted 2025-06-06; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Temporomandibular Disorders (TMD); Temporomandibular Pain; Hypermobility Syndrome (Disorder); Hypermobility, Joint; Arthrocentesis; Prolotherapy
Keywords: hypermobility; subluxation; prolotherapy; arthrocentesis
MeSH Terms: conditions — Temporomandibular Joint Disorders; Joint Instability; Joint Dislocations | interventions — Glucose; Arthrocentesis; Ringer's Solution

STUDY DESIGN:
Intervention Model Description: The first group applied prolotherapy, while the other group applied arthrocentesis and prolotherapy together.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Combined Prolotherapy Group (Experimental): Patients with TMJ hypermobility underwent arthrocentesis for joint pain in addition to prolotherapy.
  Interventions: Drug: prolotherapy solution of 20% dextrose; Drug: Arthrocentesis with ringer solution
- Traditional Prolotherapy Group (Active Comparator): Prolotherapy was applied to patients with TMJ hypermobility.
  Interventions: Drug: prolotherapy solution of 20% dextrose

INTERVENTIONS:
Drug: prolotherapy solution of 20% dextrose — Polotherapy, it involves injecting an irritant solution into weakened joints, ligaments, or tendons to stimulate collagen production and tissue repair at fibro-osseous junctions.
Drug: Arthrocentesis with ringer solution — Integrating arthrocentesis with prolotherapy may enhance therapeutic outcomes by addressing both the mechanical and inflammatory aspects of TMJ hypermobility. This dual-modality technique presents a promising minimally invasive option for clinicians managing patients with joint instability.
  Arms: Combined Prolotherapy Group

SUMMARY:
1. Diagnosis and Indication You have been diagnosed with temporomandibular joint (TMJ) hypermobility and/or dysfunction, characterized by symptoms such as jaw clicking, locking, pain in the joint area, or difficulty in opening and closing the mouth. After clinical and radiographic evaluation, the recommended treatment includes arthrocentesis and prolotherapy, either alone or in combination.
2. Description of Procedures

   A. TMJ Arthrocentesis:

   This is a minimally invasive procedure in which small needles are inserted into the TMJ space to irrigate the joint using sterile fluid (e.g., Ringer's solution). The procedure aims to eliminate inflammatory mediators, release joint adhesions, and improve mandibular mobility. It is generally performed under local anesthesia in an outpatient setting.

   B. Prolotherapy:

   Prolotherapy involves the injection of an irritant solution (typically dextrose combined with a local anesthetic) into the joint capsule, ligaments, or surrounding tissue. The goal is to stimulate the body's natural healing response, promoting collagen production and tissue regeneration to improve joint stability and function.

   C. Combined Approach:

   In certain cases, both treatments may be performed during the same session to maximize clinical benefit-arthrocentesis addresses inflammation and mobility, while prolotherapy enhances long-term stabilization.
3. Benefits and Expected Outcomes Reduction in TMJ pain and joint clicking

   Improved jaw function and range of motion

   Stabilization of the joint and reduced recurrence of dislocation or subluxation

   Minimally invasive and generally well-tolerated
4. Possible Risks and Complications

   Although these procedures are generally safe, potential risks may include but are not limited to:

   Mild pain or swelling at the injection site

   Temporary facial numbness or weakness (rare and usually self-resolving)

   Dizziness or light-headedness

   Joint stiffness or infection (very rare)

   Allergic reaction to anesthetic or injected substances
5. Alternatives to the Proposed Procedure

   You have the right to consider other treatment options, which may include:

   Physical therapy or jaw exercises

   Oral splints or bite guards

   Medication (analgesics, muscle relaxants)

   Surgical interventions (if conservative methods fail)
6. Patient Instructions and Post-Procedure Care Avoid wide mouth opening, yawning, or chewing hard foods for several days

Use only recommended medications (e.g., acetaminophen/paracetamol); avoid anti-inflammatory drugs unless advised otherwise

Apply cold compresses to reduce swelling if necessary

Attend all scheduled follow-up appointments

Notify your doctor immediately if you experience severe pain, prolonged numbness, fever, or signs of infection

ELIGIBILITY:
Inclusion Criteria:

* patients with unilateral or bilateral TMJ hypermobility
* history of open locking
* complaints of joint sounds and facial pain
* treated with combine or traditionally prolotherapy
* followed for at least 3 months
* the diagnosis of the patients was confirmed by TMJ radiography

Exclusion Criteria:

* patients who underwent discectomy
* patients with active infection (fever, redness, oedema, loss of function, etc.)
* pathological findings (tumour, cyst, etc.) in the related area were excluded
* patients with systemic disorders that could affect the results

Ages: 17 Years to 46 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Pain intensity of TMJ | From pre-treatment to the 3rd month after treatment
  Pain intensity of TMJ evaluated by visual analog scale (VAS) questionnaire. VAS is designated by an marked horizontal line, 10 mm long, scored from 0 (no pain) to 10 (intolerable pain), anchored by word identifiers at each end. Patients marked the point on the line that they thought represented their current situation.

SECONDARY OUTCOMES:
Maximal interincisal opening (MIO) | From pre-treatment to the 3rd month after treatment
  Maximal interincisal opening (MIO) was recorded by measuring the distance between the incisal edges of the upper and lower incisors in the midline with the help of a ruler. Maximal interincisal opening was measured preoperatively (T0), postoperatively 1 week (T1), 1 month (T2) and 3 months (T3).

OTHER OUTCOMES:
TMJ sounds | From pre-treatment to the 3rd month after treatment
  TMJ sounds were evaluated as click or no click during mouth opening. The presence of clicking sound and pain were evaluated preoperatively and 3 months. The other variables studied were demographic data (gender and age) and the affected side.

CONTACTS AND LOCATIONS:
Locations (1):
- Karadeniz Technical University, Trabzon, Trabzon, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 2019-2022

REFERENCES:
- [Background] Comert Kilic S, Gungormus M. Is dextrose prolotherapy superior to placebo for the treatment of temporomandibular joint hypermobility? A randomized clinical trial. Int J Oral Maxillofac Surg. 2016 Jul;45(7):813-9. doi: 10.1016/j.ijom.2016.01.006. Epub 2016 Feb 2. PMID 26846795
- [Background] Dasukil S, Shetty SK, Arora G, Degala S. Efficacy of Prolotherapy in Temporomandibular Joint Disorders: An Exploratory Study. J Maxillofac Oral Surg. 2021 Mar;20(1):115-120. doi: 10.1007/s12663-020-01328-9. Epub 2020 Jan 13. PMID 33584052
- [Background] Taskesen F, Cezairli B. Efficacy of prolotherapy and arthrocentesis in management of temporomandibular joint hypermobility. Cranio. 2023 Sep;41(5):423-431. doi: 10.1080/08869634.2020.1861887. Epub 2020 Dec 16. PMID 33326351
- [Background] Cezairli B, Sivrikaya EC, Omezli MM, Ayranci F, Seyhan Cezairli N. Results of Combined, Single-Session Arthrocentesis and Dextrose Prolotherapy for Symptomatic Temporomandibular Joint Syndrome: A Case Series. J Altern Complement Med. 2017 Oct;23(10):771-777. doi: 10.1089/acm.2017.0068. Epub 2017 Oct 10. PMID 29017019
- [Background] Abbadi W, Kara Beit Z, Al-Khanati NM. Arthrocentesis, Injectable Platelet-Rich Plasma and Combination of Both Protocols of Temporomandibular Joint Disorders Management: A Single-Blinded Randomized Clinical Trial. Cureus. 2022 Nov 11;14(11):e31396. doi: 10.7759/cureus.31396. eCollection 2022 Nov. PMID 36523721
- [Background] Dagenais S, Wooley J, Hite M, Green R, Mayer J. Acute toxicity evaluation of proliferol: a dose-escalating, placebo-controlled study in swine. Int J Toxicol. 2009 May-Jun;28(3):219-29. doi: 10.1177/1091581809336478. PMID 19546260
- [Background] Refai H. Long-term therapeutic effects of dextrose prolotherapy in patients with hypermobility of the temporomandibular joint: a single-arm study with 1-4 years' follow up. Br J Oral Maxillofac Surg. 2017 Jun;55(5):465-470. doi: 10.1016/j.bjoms.2016.12.002. Epub 2017 Apr 29. PMID 28460873
- [Background] Gibaly A, Abdelmoiz M, Alghandour AN. Evaluation of the effect of dextrose prolotherapy versus deep dry needling therapy for the treatment of temporomandibular joint anterior disc displacement with reduction: (a randomized controlled trial). Clin Oral Investig. 2024 Aug 8;28(9):475. doi: 10.1007/s00784-024-05830-z. PMID 39115583
- [Background] Zhou H, Hu K, Ding Y. Modified dextrose prolotherapy for recurrent temporomandibular joint dislocation. Br J Oral Maxillofac Surg. 2014 Jan;52(1):63-6. doi: 10.1016/j.bjoms.2013.08.018. Epub 2013 Sep 21. PMID 24064304
- [Background] Ungor C, Atasoy KT, Taskesen F, Cezairli B, Dayisoylu EH, Tosun E, Senel FC. Short-term results of prolotherapy in the management of temporomandibular joint dislocation. J Craniofac Surg. 2013 Mar;24(2):411-5. doi: 10.1097/SCS.0b013e31827ff14f. PMID 23524704
- [Background] Nagori SA, Jose A, Gopalakrishnan V, Roy ID, Chattopadhyay PK, Roychoudhury A. The efficacy of dextrose prolotherapy over placebo for temporomandibular joint hypermobility: A systematic review and meta-analysis. J Oral Rehabil. 2018 Dec;45(12):998-1006. doi: 10.1111/joor.12698. Epub 2018 Aug 3. PMID 30024045
- [Background] Foster TE, Puskas BL, Mandelbaum BR, Gerhardt MB, Rodeo SA. Platelet-rich plasma: from basic science to clinical applications. Am J Sports Med. 2009 Nov;37(11):2259-72. doi: 10.1177/0363546509349921. PMID 19875361
- [Background] Distel LM, Best TM. Prolotherapy: a clinical review of its role in treating chronic musculoskeletal pain. PM R. 2011 Jun;3(6 Suppl 1):S78-81. doi: 10.1016/j.pmrj.2011.04.003. PMID 21703585
- [Background] Nitzan DW, Dolwick MF, Martinez GA. Temporomandibular joint arthrocentesis: a simplified treatment for severe, limited mouth opening. J Oral Maxillofac Surg. 1991 Nov;49(11):1163-7; discussion 1168-70. doi: 10.1016/0278-2391(91)90409-f. PMID 1941330
- [Background] Rabago D, Slattengren A, Zgierska A. Prolotherapy in primary care practice. Prim Care. 2010 Mar;37(1):65-80. doi: 10.1016/j.pop.2009.09.013. PMID 20188998
- [Background] Mustafa R, Gungormus M, Mollaoglu N. Evaluation of the Efficacy of Different Concentrations of Dextrose Prolotherapy in Temporomandibular Joint Hypermobility Treatment. J Craniofac Surg. 2018 Jul;29(5):e461-e465. doi: 10.1097/SCS.0000000000004480. PMID 29533255
- [Background] de Farias JF, Melo SL, Bento PM, Oliveira LS, Campos PS, de Melo DP. Correlation between temporomandibular joint morphology and disc displacement by MRI. Dentomaxillofac Radiol. 2015;44(7):20150023. doi: 10.1259/dmfr.20150023. Epub 2015 Mar 25. PMID 25806865
- [Background] Majumdar SK, Krishna S, Chatterjee A, Chakraborty R, Ansari N. Single Injection Technique Prolotherapy for Hypermobility Disorders of TMJ Using 25 % Dextrose: A Clinical Study. J Maxillofac Oral Surg. 2017 Jun;16(2):226-230. doi: 10.1007/s12663-016-0944-0. Epub 2016 Jul 25. PMID 28439165
- [Background] Refai H, Altahhan O, Elsharkawy R. The efficacy of dextrose prolotherapy for temporomandibular joint hypermobility: a preliminary prospective, randomized, double-blind, placebo-controlled clinical trial. J Oral Maxillofac Surg. 2011 Dec;69(12):2962-70. doi: 10.1016/j.joms.2011.02.128. Epub 2011 Jul 16. PMID 21757278
- [Background] Torres DE, McCain JP. Arthroscopic electrothermal capsulorrhaphy for the treatment of recurrent temporomandibular joint dislocation. Int J Oral Maxillofac Surg. 2012 Jun;41(6):681-9. doi: 10.1016/j.ijom.2012.03.008. Epub 2012 Apr 7. PMID 22487806
- [Derived] Ates H, Sivrikaya EC. Is the combine prolotherapy more effective than the traditional prolotherapy in patients with temporomandibular joint hypermobility? J Craniomaxillofac Surg. 2025 Dec;53(12):2238-2244. doi: 10.1016/j.jcms.2025.10.008. Epub 2025 Nov 3. PMID 41188164